CLINICAL TRIAL: NCT02902419
Title: The Effect of Timing of Removal of Wound Dressing on Surgical Site Infection Rate After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Peter R Cole, MD, MD, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AlbanyMC2984
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Wound dressing removal was performed between 12-30 hours postoperatively.
  Interventions: Other: Wound dressing removal.
- 2 (Active Comparator): Wound dressing removal was performed between 30-48 hours postoperatively.
  Interventions: Other: Wound dressing removal.

INTERVENTIONS:
Other: Wound dressing removal.

SUMMARY:
A randomized controlled trial measuring surgical site infection rate as a function of timing of wound dressing removal.

DETAILED DESCRIPTION:
A randomized controlled trial with a sample size of 602 patients to study the effect of timing of wound dressing removal on the surgical site infection rate. 300 patients were randomized to a group that had the wound dressing removed between 12-30 hours postoperatively. 302 patients were randomized to a group that had the wound dressing removal between 30-48 hours postoperatively. Statistical analyses were performed to determine if the timing of dressing removal had statistical significance on the surgical site infection rate, the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients ages 18-50 years;
* medically competent (no proxies or prisoners); and
* multifetal and singleton gestations from 23 0/7 weeks to 42 0/7 weeks gestational age.

Exclusion Criteria:

* Inability to obtain informed consent;
* fetal death;
* immunocompromised patients; patients taking immuno-suppressants; history of documented surgical site infection; or patients requiring reoperation within the 6 week postoperative period for indications other than wound dehiscence/debridement/infection.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 602 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Surgical Site infection Rate | 6 weeks postoperatively
  Cellulitis, purulent drainage, abscess or wound requiring drainage, debridement, and antibiotics associated with a clinical diagnosis of infection. Any disruption of fascia or subcutaneous skin.

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Cole, MD, Principal Investigator — Albany Medical College; Kevin C Kiley, MD, Study Chair — Albany Medical College
Locations (2):
- United States (2):
  - St. Peter's Hospital, Albany, New York
  - Bellevue Women's Center, Niskayuna, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Kirmeyer S, Mathews TJ, Wilson EC. Births: final data for 2009. Natl Vital Stat Rep. 2011 Nov 3;60(1):1-70. PMID 22670489
- [Background] Poulsen KB, Bremmelgaard A, Sorensen AI, Raahave D, Petersen JV. Estimated costs of postoperative wound infections. A case-control study of marginal hospital and social security costs. Epidemiol Infect. 1994 Oct;113(2):283-95. doi: 10.1017/s0950268800051712. PMID 7925666
- [Background] Consensus paper on the surveillance of surgical wound infections. The Society for Hospital Epidemiology of America; The Association for Practitioners in Infection Control; The Centers for Disease Control; The Surgical Infection Society. Infect Control Hosp Epidemiol. 1992 Oct;13(10):599-605. PMID 1334987
- [Background] Owen J, Andrews WW. Wound complications after cesarean sections. Clin Obstet Gynecol. 1994 Dec;37(4):842-55. doi: 10.1097/00003081-199412000-00009. No abstract available. PMID 7842552
- [Background] Olsen MA, Butler AM, Willers DM, Devkota P, Gross GA, Fraser VJ. Risk factors for surgical site infection after low transverse cesarean section. Infect Control Hosp Epidemiol. 2008 Jun;29(6):477-84; discussion 485-6. doi: 10.1086/587810. PMID 18510455
- [Background] van Ramshorst GH, Nieuwenhuizen J, Hop WC, Arends P, Boom J, Jeekel J, Lange JF. Abdominal wound dehiscence in adults: development and validation of a risk model. World J Surg. 2010 Jan;34(1):20-7. doi: 10.1007/s00268-009-0277-y. PMID 19898894
- [Background] Pavlidis TE, Galatianos IN, Papaziogas BT, Lazaridis CN, Atmatzidis KS, Makris JG, Papaziogas TB. Complete dehiscence of the abdominal wound and incriminating factors. Eur J Surg. 2001 May;167(5):351-4; discussion 355. doi: 10.1080/110241501750215221. PMID 11419550
- [Background] Ovington LG. Hanging wet-to-dry dressings out to dry. Home Healthc Nurse. 2001 Aug;19(8):477-83; quiz 484. doi: 10.1097/00004045-200108000-00007. PMID 11982183
- [Background] Chen WY, Rogers AA, Lydon MJ. Characterization of biologic properties of wound fluid collected during early stages of wound healing. J Invest Dermatol. 1992 Nov;99(5):559-64. doi: 10.1111/1523-1747.ep12667378. PMID 1431216
- [Background] Toon CD, Ramamoorthy R, Davidson BR, Gurusamy KS. Early versus delayed dressing removal after primary closure of clean and clean-contaminated surgical wounds. Cochrane Database Syst Rev. 2013 Sep 5;(9):CD010259. doi: 10.1002/14651858.CD010259.pub2. PMID 24009067
- [Background] Figueroa D, Jauk VC, Szychowski JM, Garner R, Biggio JR, Andrews WW, Hauth J, Tita AT. Surgical staples compared with subcuticular suture for skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Jan;121(1):33-8. doi: 10.1097/aog.0b013e31827a072c. PMID 23262925
- [Background] Tuuli MG, Rampersad RM, Carbone JF, Stamilio D, Macones GA, Odibo AO. Staples compared with subcuticular suture for skin closure after cesarean delivery: a systematic review and meta-analysis. Obstet Gynecol. 2011 Mar;117(3):682-690. doi: 10.1097/AOG.0b013e31820ad61e. PMID 21343772
- [Background] Anderson DJ, Podgorny K, Berrios-Torres SI, Bratzler DW, Dellinger EP, Greene L, Nyquist AC, Saiman L, Yokoe DS, Maragakis LL, Kaye KS. Strategies to prevent surgical site infections in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Jun;35(6):605-27. doi: 10.1086/676022. PMID 24799638